CLINICAL TRIAL: NCT00932217
Title: Study on the Incidence of Febrile Episodes During Stem Cells Collection After Chemotherapy in Patients With Multiple Myeloma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Pisa (Other)
Responsible Party: Mario Petrini, University of Pisa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Pisa 01
Record Dates: First submitted 2009-07-02; First posted 2009-07-03 (Estimated); Last update posted 2009-07-03 (Estimated); Status verified 2009-02

CONDITIONS: G-CSF, Multiple Myeloma, Febrile Episode, Filgrastim, Leograstim
MeSH Terms: conditions — Multiple Myeloma | interventions — Filgrastim; Lenograstim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- filgrastim (Active Comparator): patients mobilized with filgrastim
  Interventions: Drug: filgrastim
- lenograstim (Active Comparator): patients mobilized with lenograstim
  Interventions: Drug: lenograstim

INTERVENTIONS:
Drug: filgrastim — subcutaneous filgrastim administration
  Arms: filgrastim
Drug: lenograstim — subcutaneous lenograstim administration
  Arms: lenograstim

SUMMARY:
To evaluate the difference in the incidence of febrile episodes in patients undergoing stem cells mobilization with chemotherapy and filgrastim versus chemotherapy and lenograstim.

A febrile episode will be considered as: body temperature > 38°C for two measurements in the 24 hours with an interval of 6 hours at least between the two measurements.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 and < 70 years
2. Diagnosis of multiple myeloma
3. ECOG < 2 to be evaluated at baseline, after the induction chemotherapy
4. Indication to the mobilization with high dose cyclophosphamide chemotherapy
5. Normal blood counts: neutrophils > 1500/μl; platelets > 100.000/μl; hemoglobin > 10 g/dl.
6. Liver and renal function: SGOT/AST, SGPT/ALT; bilirubin < 1.5 times the upper limit of the normal ranges; creatinine < 2 times the upper limit of the normal ranges.
7. Interval from previous induction chemotherapy to high dose chemotherapy between 30 and 60 days
8. ECG e/o Echocardiogram within age related normal range
9. Negative HCV and HbsAg
10. Must be willing and able to fill in the patient's diary
11. Written informed consent

Exclusion Criteria:

1. Documented and/or suspected infections
2. Uncontrolled concurrent illness
3. Documented cardiac dysfunction

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2004-12; Primary Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
febrile episode | 30 days

SECONDARY OUTCOMES:
Documented infectious episodes Collection efficiency (CD34+ cells/kilo) Mobilization days Safety | 30 days

REFERENCES:
- [Background] Layton JE, Hall NE. The interaction of G-CSF with its receptor. Front Biosci. 2006 Sep 1;11:3181-9. doi: 10.2741/2041. PMID 16720384
- [Background] Martin-Christin F. Granulocyte colony stimulating factors: how different are they? How to make a decision? Anticancer Drugs. 2001 Mar;12(3):185-91. doi: 10.1097/00001813-200103000-00002. PMID 11290864
- [Background] Ono M. Physicochemical and biochemical characteristics of glycosylated recombinant human granulocyte colony stimulating factor (lenograstim). Eur J Cancer. 1994;30A Suppl 3:S7-11. PMID 7535073
- [Background] Carter CR, Whitmore KM, Thorpe R. The significance of carbohydrates on G-CSF: differential sensitivity of G-CSFs to human neutrophil elastase degradation. J Leukoc Biol. 2004 Mar;75(3):515-22. doi: 10.1189/jlb.0803378. Epub 2003 Dec 4. PMID 14657210
- [Background] Oh-eda M, Hasegawa M, Hattori K, Kuboniwa H, Kojima T, Orita T, Tomonou K, Yamazaki T, Ochi N. O-linked sugar chain of human granulocyte colony-stimulating factor protects it against polymerization and denaturation allowing it to retain its biological activity. J Biol Chem. 1990 Jul 15;265(20):11432-5. PMID 1694845
- [Background] Watts MJ, Addison I, Long SG, Hartley S, Warrington S, Boyce M, Linch DC. Crossover study of the haematological effects and pharmacokinetics of glycosylated and non-glycosylated G-CSF in healthy volunteers. Br J Haematol. 1997 Aug;98(2):474-9. doi: 10.1046/j.1365-2141.1997.2393053.x. PMID 9266953
- [Background] Molineux G. The design and development of pegfilgrastim (PEG-rmetHuG-CSF, Neulasta). Curr Pharm Des. 2004;10(11):1235-44. doi: 10.2174/1381612043452613. PMID 15078138
- [Background] Mattii L, Azzara A, Fazzi R, Carulli G, Chimenti M, Cecconi N, Galimberti S, Petrini M. Glycosylated or non-glycosylated G-CSF differently influence human granulocyte functions through RhoA. Leuk Res. 2005 Nov;29(11):1285-92. doi: 10.1016/j.leukres.2005.04.011. PMID 15916805
- [Background] Azzara A, Carulli G, Rizzuti-Gullaci A, Capochiani E, Petrini M. Lenograstim and filgrastim effects on neutrophil motility in patients undergoing chemotherapy: evaluation by computer-assisted image analysis. Am J Hematol. 2001 Apr;66(4):306-7. doi: 10.1002/ajh.1064. No abstract available. PMID 11279646
- [Background] Ribeiro D, Veldwijk MR, Benner A, Laufs S, Wenz F, Ho AD, Fruehauf S. Differences in functional activity and antigen expression of granulocytes primed in vivo with filgrastim, lenograstim, or pegfilgrastim. Transfusion. 2007 Jun;47(6):969-80. doi: 10.1111/j.1537-2995.2007.01241.x. PMID 17524085
- [Background] Bodey GP, Buckley M, Sathe YS, Freireich EJ. Quantitative relationships between circulating leukocytes and infection in patients with acute leukemia. Ann Intern Med. 1966 Feb;64(2):328-40. doi: 10.7326/0003-4819-64-2-328. No abstract available. PMID 5216294
- [Background] Clark OA, Lyman GH, Castro AA, Clark LG, Djulbegovic B. Colony-stimulating factors for chemotherapy-induced febrile neutropenia: a meta-analysis of randomized controlled trials. J Clin Oncol. 2005 Jun 20;23(18):4198-214. doi: 10.1200/JCO.2005.05.645. PMID 15961767
- [Background] Trillet-Lenoir V, Green J, Manegold C, Von Pawel J, Gatzemeier U, Lebeau B, Depierre A, Johnson P, Decoster G, Tomita D, et al. Recombinant granulocyte colony stimulating factor reduces the infectious complications of cytotoxic chemotherapy. Eur J Cancer. 1993;29A(3):319-24. doi: 10.1016/0959-8049(93)90376-q. PMID 7691119
- [Background] Green MD, Koelbl H, Baselga J, Galid A, Guillem V, Gascon P, Siena S, Lalisang RI, Samonigg H, Clemens MR, Zani V, Liang BC, Renwick J, Piccart MJ; International Pegfilgrastim 749 Study Group. A randomized double-blind multicenter phase III study of fixed-dose single-administration pegfilgrastim versus daily filgrastim in patients receiving myelosuppressive chemotherapy. Ann Oncol. 2003 Jan;14(1):29-35. doi: 10.1093/annonc/mdg019. PMID 12488289
- [Background] Hoglund M, Smedmyr B, Bengtsson M, Totterman TH, Cour-Chabernaud V, Yver A, Simonsson B. Mobilization of CD34+ cells by glycosylated and nonglycosylated G-CSF in healthy volunteers--a comparative study. Eur J Haematol. 1997 Sep;59(3):177-83. doi: 10.1111/j.1600-0609.1997.tb00972.x. PMID 9310126
- [Background] de Arriba F, Lozano ML, Ortuno F, Heras I, Moraleda JM, Vicente V. Prospective randomized study comparing the efficacy of bioequivalent doses of glycosylated and nonglycosylated rG-CSF for mobilizing peripheral blood progenitor cells. Br J Haematol. 1997 Feb;96(2):418-20. doi: 10.1046/j.1365-2141.1997.d01-2029.x. PMID 9029036
- [Background] Ings SJ, Balsa C, Leverett D, Mackinnon S, Linch DC, Watts MJ. Peripheral blood stem cell yield in 400 normal donors mobilised with granulocyte colony-stimulating factor (G-CSF): impact of age, sex, donor weight and type of G-CSF used. Br J Haematol. 2006 Sep;134(5):517-25. doi: 10.1111/j.1365-2141.2006.06223.x. PMID 17018030
- [Background] Fischer JC, Frick M, Wassmuth R, Platz A, Punzel M, Wernet P. Superior mobilisation of haematopoietic progenitor cells with glycosylated G-CSF in male but not female unrelated stem cell donors. Br J Haematol. 2005 Sep;130(5):740-6. doi: 10.1111/j.1365-2141.2005.05678.x. PMID 16115131